CLINICAL TRIAL: NCT02049216
Title: The Effect of Flexible Tape Versus Placebo Tape in Patients Completing a Home Exercise Program With Knee Osteoarthritis
Brief Title: The Effect of Flexible Tape in Knee Osteoarthritis
Acronym: FTKOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Alfred (Other)
Responsible Party: Principal Investigator, Kim McManus, Physiotherapist, The Alfred
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FTKOA
Record Dates: First submitted 2014-01-22; First posted 2014-01-30 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Osteoarthritis
Keywords: knee; osteoarthritis; tape; exercise; rocktape
MeSH Terms: conditions — Osteoarthritis; Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham tape (Sham Comparator): * Fixomull tape only
  * Single piece of 10cm wide, 32cm long applied from inferior to tibial tuberosity, over patella and onto quadriceps muscle. Corners rounded. Tape to be applied with the knee in 90 degrees flexion.
  Participants in both groups will also be prescribed an individualised home exercise program by a physiotherapist.
  Interventions: Other: Fixomull; Other: Exercise
- Flexible tape (Experimental): Flexible tape (rocktape brand) applied as follows:
  First piece of tape 10 cm wide and 32cm long (length of a standard goniometer). Split down centre 18cm from 1 end. Second piece of tape 5cm wide and 14cm long.
  Tape applied in 90 degrees knee flexion Applied with no tension in proximal and distal ends. 30% tension to un-split portion placed over quads. 50% tension to split portion placed either side of patella and crossing over at tibial tuberosity Additional piece of 5cm wide flexible tape applied with 80% tension over patella tendon, with no tension in 3cm from ends All tape corners rounded
  Participants in both groups will also be prescribed an individualised home exercise program by a physiotherapist.
  Interventions: Other: Flexible tape; Other: Exercise

INTERVENTIONS:
Other: Flexible tape — Flexible, elasticised, adhesive athletic tape
  Other Names: Rocktape
  Arms: Flexible tape
Other: Fixomull
  Other Names: Hypa fix; Medical adhesive tape
  Arms: Sham tape
Other: Exercise — Participants in both groups will be prescribed a home exercise program to complete.
  Other Names: Strengthening

SUMMARY:
People with osteoarthritis (OA) of the knee attending The Alfred hospital will be invited to participate in a randomised controlled trial comparing two different types of knee taping. Both groups will also be prescribed an exercise program to assist in management of their knee OA.

Hypothesis are as follows:

1. Participants treated with flexible tape with have greater reductions in pain and improvements on timed performance based measures when compared to those treated with a placebo tape.
2. Participants in both groups will have clinically significant improvements in pain and timed performance based measures compared to their baseline scores.

DETAILED DESCRIPTION:
Interventions:

Participants in both groups will attend physiotherapy on 4 occasions, in addition to an initial appointment where baseline data will be collected.

All participants will be provided with an individualised home exercise program. This will be provided based on the investigators' clinical experience and evidence based programs. The participant will be provided with a handout detailing the exercises they are to complete, including dosage. If there is excessive pain or difficulty associated with completing an exercise the participant will be advised to cease that particular exercise until they have been reviewed by the researcher the following week.

Participants will have their knee taped according to either the therapeutic flexible taping protocol, or the placebo taping protocol depending on which group they have been randomly allocated to on three occasions at one week intervals. All participants will be provided with written information regarding tape allergies and when to remove the tape from their knee. To control for the Hawthorne effect participants will not be aware of whether they are in the intervention or placebo group.

Participants will attend for appointments once per week for three weeks. They will then have a three week period of no intervention and return for a review and completion of the study. At this time the participant can be referred for further physiotherapy intervention as is clinically indicated. This may include physiotherapy at The Alfred Hospital, private practice or the participants' local health services.

If at anytime a participant wishes to withdraw from the study they can be referred by the investigators to continue their physiotherapy in the appropriate setting.

Sample size calculations: The investigators hypothesise that the combination of taping and an exercise program will give rise to clinically significant improvements in functional capacity, symptoms and quality of life. If there is truly no difference in the change in VAS between placebo and therapeutic based groups, then 30 patients are required to be 90% sure that the 95% confidence interval will exclude a difference in means of more than 20mm. This has been demonstrated by Tubach and colleagues in 2005. This assumes a standard deviation of the change in VAS of 21.5. Due to participant attrition anticipated an additional 20% will be recruited to the sample. This will total 36 participants in total.

Feasibility: The osteoarthritis hip and knee clinic at The Alfred hospital review approximately 13 patients per week of which the majority would be appropriate for inclusion in this trial. There are also many referrals from orthopaedics, rheumatology and emergency for patients who will be appropriate for inclusion. It is therefore anticipated that recruitment to the study will not be a barrier to completion of this trial.

Statistical analysis: All data will be analysed by intention to treat. Continuous variables will be analysed using analysis of covariance, controlling for baseline values and recruitment centre. The proportion of participants who complete the program will be compared between groups using a chi-squared test and the relative risk of non-completion will be determined. Alpha will be set at 0.05

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of osteoarthritis of the knee
* radiological diagnosis of osteoarthritis of the knee
* able to understand basic English
* knee outcome and injury scale available in patients's preferred language

Exclusion Criteria:

* other significant lower limb pathology
* previous total knee replacement in effected knee
* co-morbidities limiting participation in a basic home exercise program or performance of outcome measures eg. unstable cardiac or respiratory conditions

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in pain on visual analogue scale | baseline, 0,3 and 6 weeks after commencement of intervention
  • Pain on a Visual Analogue Scale (VAS) over last 48hrs at rest and movement. Anchors used will be no pain and worst imaginable pain. The VAS has been found to be valid, reliable and sensitive to change in this population (Tubach et al, 2005)

SECONDARY OUTCOMES:
Chang in Knee injury and osteoarthritis outcome score (excluding sport domain) | baseline, one week, three weeks and six weeks
  The KOOS, a valid and reliable functional questionnaire in patients with knee conditions covering the domains of function, symptoms, quality of life and sport . Sport will not be included in analysis as this is not relevant to the study population.

OTHER OUTCOMES:
Change in 30 sec STS test | baseline, 1 week from baseline with no intervention (control period), immediately after the first tape application (one week), three weeks and six weeks
  The maximum number of chair stand repetitions possible in a 30 second period as per protocol available at:
  http://www.oarsi.org/sites/default/files/docs/2013/manual.pdf
Change in time taken to climb 3 steps | baseline, 1 week from baseline with no intervention (control period), immediately after the first tape application (one week), three weeks and six weeks
  The time (in seconds) it takes to ascend and descend a 3 stairs as per protocol available at:
  http://www.oarsi.org/sites/default/files/docs/2013/manual.pdf
Change in time to complete 40m walk test | baseline, 1 week from baseline with no intervention (control period), immediately after the first tape application (one week), three weeks and six weeks
  A fast-paced walking test that is timed over 4 x 10m (33 ft) for a total 40 m (132 ft) as per protocol available at:
  http://www.oarsi.org/sites/default/files/docs/2013/manual.pdf
Change in pain on visual analogue scale (VAS) during 30 sec sit to stand test | prior to initial knee taping and 30mins later following knee tape
  Once 30sec sit to stand is completed participants to rate pain on VAS
Change in pain on visual analogue scale (VAS) 40m walk test | prior to initial knee taping and 30mins later following knee tape
  Once 40m walk test is completed participants to rate pain on VAS
Change in pain on visual analogue scale (VAS) 3 stair climb test | prior to initial knee taping and 30mins later following knee tape
  Once 3 stair climb test is completed participants to rate pain on VAS
Change in amount of weekly analgesia medication consumed | weekly for 4 weeks
  Participants will be asked to keep a record of the number of tablets they take per week for pain relief. This will be compared within each particiapnt over the first four weeks of the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Kim L McManus, B, Physio, Principal Investigator — The Alfred
Locations (1):
- The Alfred Hospital, Prahran, Victoria, Australia

REFERENCES:
- [Background] Tubach F, Ravaud P, Baron G, Falissard B, Logeart I, Bellamy N, Bombardier C, Felson D, Hochberg M, van der Heijde D, Dougados M. Evaluation of clinically relevant changes in patient reported outcomes in knee and hip osteoarthritis: the minimal clinically important improvement. Ann Rheum Dis. 2005 Jan;64(1):29-33. doi: 10.1136/ard.2004.022905. Epub 2004 Jun 18. PMID 15208174
- [Background] Bennell KL, Hinman RS. A review of the clinical evidence for exercise in osteoarthritis of the hip and knee. J Sci Med Sport. 2011 Jan;14(1):4-9. doi: 10.1016/j.jsams.2010.08.002. Epub 2010 Sep 17. PMID 20851051
- [Derived] McManus KL, Kimmel LA, Holland AE. Rocktape provides no benefit over sham taping in people with knee osteoarthritis who are completing an exercise program: a randomised trial. Physiotherapy. 2021 Dec;113:29-36. doi: 10.1016/j.physio.2021.05.005. Epub 2021 May 17. PMID 34555671